CLINICAL TRIAL: NCT04084808
Title: Ingestion of Maple Products During High Intensity Intermittent Exercise : Effects on Cognitive Flexibility
Brief Title: Maple Products and Cognitive Performance During High Intensity Intermittent Exercise (HIIE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Fédération des producteurs acéricoles du Québec (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Maple-cognition-exercise
Record Dates: First submitted 2019-08-20; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Carbohydrate Ingestion; Cognitive Performance; High Intensity Interval Training
MeSH Terms: interventions — Blood Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Maple Syrup (Experimental): A maple syrup solution of 6% carbohydrate per volume labeled with 13C-sucrose will first be ingested at rest (167 mL), right before starting warmup. Another dose (167 mL) will be administered after warmup. Four additional doses of 167 mL will be ingested immediately after the first four 3-minute bouts at 95% of Maximal Aerobic Power. A final dose (167 mL) will be ingested after the last effort.
  Interventions: Dietary Supplement: Solution ingestion; Behavioral: Cognitive flexibility; Procedure: Brain oxygenation; Other: Palatability; Procedure: Blood glucose; Behavioral: Perceived exertion; Behavioral: High Intensity Interval Training bouts
- Maple sap (Experimental): A maple sap solution of 6% carbohydrate per volume labeled with 13C-sucrose will first be ingested at rest (167 mL), right before starting warmup. Another dose (167 mL) will be administered after warmup. Four additional doses of 167 mL will be ingested immediately after the first four 3-minute bouts at 95% of Maximal Aerobic Power. A final dose (167 mL) will be ingested after the last effort.
  Interventions: Dietary Supplement: Solution ingestion; Behavioral: Cognitive flexibility; Procedure: Brain oxygenation; Other: Palatability; Procedure: Blood glucose; Behavioral: Perceived exertion; Behavioral: High Intensity Interval Training bouts
- Glucose (Active Comparator): A glucose solution of 6% carbohydrate per volume labeled with 13C-sucrose will first be ingested at rest (167 mL), right before starting warmup. Another dose (167 mL) will be administered after warmup. Four additional doses of 167 mL will be ingested immediately after the first four 3-minute bouts at 95% of Maximal Aerobic Power. A final dose (167 mL) will be ingested after the last effort.
  Interventions: Dietary Supplement: Solution ingestion; Behavioral: Cognitive flexibility; Procedure: Brain oxygenation; Other: Palatability; Procedure: Blood glucose; Behavioral: Perceived exertion; Behavioral: High Intensity Interval Training bouts
- Sports drink (Active Comparator): A commercial sports drink of 6% carbohydrate per volume labeled with 13C-sucrose will first be ingested at rest (167 mL), right before starting warmup. Another dose (167 mL) will be administered after warmup. Four additional doses of 167 mL will be ingested immediately after the first four 3-minute bouts at 95% of Maximal Aerobic Power. A final dose (167 mL) will be ingested after the last effort.
  Interventions: Dietary Supplement: Solution ingestion; Behavioral: Cognitive flexibility; Procedure: Brain oxygenation; Other: Palatability; Procedure: Blood glucose; Behavioral: Perceived exertion; Behavioral: High Intensity Interval Training bouts
- Water (Placebo Comparator): A solution containing stevia (sugar substitute) labeled with 13C-sucrose will first be ingested at rest (167 mL), right before starting warmup. Another dose (167 mL) will be administered after warmup. Four additional doses of 167 mL will be ingested immediately after the first four 3-minute bouts at 95% of Maximal Aerobic Power. A final dose (167 mL) will be ingested after the last effort.
  Interventions: Dietary Supplement: Solution ingestion; Behavioral: Cognitive flexibility; Procedure: Brain oxygenation; Other: Palatability; Procedure: Blood glucose; Behavioral: Perceived exertion; Behavioral: High Intensity Interval Training bouts

INTERVENTIONS:
Dietary Supplement: Solution ingestion — Subjects will be required to ingest 1 liter of the experimental solution, spread over the 45 minutes of exercise. A first ingestion of 167 mL of solution will be made at rest, right before starting warmup, and another dose (167 mL) after it. Four additional doses of 167 mL will be ingested immediately after the first four 3-minute bouts at 95% of Maximal Aerobic Power. A final dose (167 mL) will be ingested after the last effort.
Behavioral: Cognitive flexibility — Subjects will be required to undergo the Stroop task. They will have to answer as quickly as possible, with push buttons, to a colour stimulus, following specific rules, and get the highest possible number of right answers. The flexibility block will show a pre-signal on a screen in front of the subject (a square or a cross will be shown). The form presented will indicate if the subject must use the colour of the writing, or the word written. Each block will consist of 50 trials, 25% of which switching the condition of answer. During this test, reaction time in milliseconds (ms) as well as the number of right answers will be measured.
  This test will be measured before the exercise protocol, during the 3-minutes exercise bouts, and every 15 minutes during the 45 minutes following exercise.
Procedure: Brain oxygenation — Optic imagery (Near-infrared spectroscopy, or NIRS) is a non-invasive technique allowing a fine investigation of the inner workings of the brain. It allows discrimination of oxygenated hemoglobin from deoxygenated hemoglobin, which informs on the coupling between blood flow and oxygen consumption inside the brain. To measure brain oxygenation with NIRS, optodes will be installed on the subject's skin without glue or transmission gel.
  [ Time Frame: During Stroop's task (i.e.before the exercise protocol, during the 3-minutes exercise bouts, and every 15 minutes during the 45 minutes following exercise). ] Measured with near-infrared spectroscopy (NIRS).
Other: Palatability — Subjects will be asked to fill out a short form on the palatability of the solution ingestion, after ingesting the first solution and at the end of exercise, after ingestion the last solution.
Procedure: Blood glucose — Blood glucose will be measured with a puncture on the tip of a finger to get a droplet of blood.
Behavioral: Perceived exertion — Perceived exertion will be assessed using 3 scales : Borg (RPE), and DP-15 scale for mental effort (Delignières, Brisswalter, & Legros, 1994). These scales will be administrated at the end of each 3 minute high intensity bout.
Behavioral: High Intensity Interval Training bouts — 6 3-minute bouts at 95% of maximal aerobic power will be done on a bike. Each bout will be separated by 3 minutes of passive recovery. The last bout will be followed by 45 minutes of rest.

SUMMARY:
The purpose of this study is to compare the cognitive performance following the ingestion of carbohydrate solutions containing either maple syrup, maple sap, corn syrup, a commercial sport drink or water.

DETAILED DESCRIPTION:
The study will require 4 meetings for each subject: a 30-minute meeting to explain the project; a meeting of 2 hours (glucose tolerance test, at rest); a one-hour meeting (maximum oxygen consumption test (VO2max) during an exercise conducted on an electromagnetically braked cycle ergometer, and a meeting of about 1,5 hours for experimentation (warmup, and 6 X 3-minutes intermittent efforts at 95% of MAP on a stationary bicycle with ingestion of a solution carbohydrates or sweetened water).

Visit #1 - Pre-participation (screening visit) Following an initial contact by phone or email, the subject will be invited to individual meetings which will last about 15 minutes. During the meeting, one of the project managers will check the eligibility of the potential subject in the study and, if eligible, will present him the details of the protocol specifying the discomforts and risks involved. The participant will be required to fill a Physical Activity Readiness Questionnaire (PAR-Q) and will be given a copy of the consent form. We will request the name and contact details of a person to contact in case of emergency, this information will be recorded and preserved in the subject matter. A period of at least three days will be allocated to make the decision whether to participate in the study or not. If the participant decides to participate in the study, he will be invited for the second visit (oral glucose tolerance test) and on this occasion will sign the consent form.

Visit #2 - Oral glucose tolerance test (OGTT) This test will be performed at Exercise Physiology Laboratory at the Department of kinesiology from the University of Montreal under the procedure commonly used for these tests. This procedure requires the ingestion of 300 mL of water containing 75 g of glucose in the morning (around 8am) after 12 hours of fasting, and blood samples and on the tip of a finger at 0, 60 and 120 minutes for the measurement of blood glucose. Subjects with higher blood glucose than 5 mmol/L before ingestion of glucose and greater than 8 mmol/L after ingestion (60 or 120 min) will not be considered for the study. These glucose tolerance standards are more stringent than those of the World Health Organization, because the objective of this test is not a diagnosis on glucose tolerance or a prognosis of its future development, but just n include in the study subjects who have good glucose tolerance.

Visit #3 - Maximum oxygen uptake testing: cycling VO2max This test will be conducted in the Exercise Physiology Laboratory at the Department of kinesiology from the University of Montreal. Exercise involves pedaling a stationary bike at a power output (resistance) gradually increasing until reaching VO2max. During the execution of the test, the subject is wearing surface electrodes to measure heart rate, a mouthpiece and nose clip to measure the volume of expired gas as well as the oxygen and carbon dioxide content to determine the consumption oxygen and carbon dioxide production. This type of testing is routinely used in our laboratory. The test can be stopped at any time by the will of the subject. For this test, guidelines established by the Exercise Physiology Laboratory at the Department of kinesiology from the University of Montreal will be followed. These guidelines are based on recommendations of ethics and safety of the "American College of Sports Medicine".

Visit #4 - Experimentation: The tests will be conducted at the Exercise Physiology Laboratory at the Department of kinesiology from the University of Montreal. The exercise is carried out on stationary cycle ergometer. Prior to exercise, electrodes (EMG) will be installed on the subject's hands, optodes helmet (NIRS) will be installed on the subject's head, and a first dose (167 mL) of a solution of carbohydrates, (120 g, 6% carbohydrate by volume), sweetened or unsweetened water will be administrated to the subject. During exercise protocol, the following solutions will be administered to the subject in a balanced, randomized, double-blind model: maple sap, maple syrup, glucose, a commercial sports drink and water. He will then begin a standardized warmup consisting of 10 minutes cycling at 40% of MAP followed by 6 bouts of 10 seconds at 95% of MAP separated by 50 seconds of passive recovery. After the second dose of solution (167 mL), the subject will have to do 6 efforts of 3 minutes at 95% of MAP, each bout separated by 3 minutes of passive recovery. He will be administered an additional dose after the first 4 efforts (4 X 167 mL). After the last effort, one last dose (167 mL) will be administered, and the subject will be asked to stay in the laboratory for the 45 minutes following the last effort. Cognitive task as well as blood sugar level will be evaluated before the exercise protocol, during the 3-minutes exercise bouts, and every 15 minutes during the 45 minutes following exercise. Heart rate, brain oxidation and muscle electrical activity will be measured continuously during recovery. The total duration of this visit is approximately 90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Low alcohol consumption (<3 drinks/week)
* Not regularly taking medication for a known pathology
* Regularly practices endurance sports (cycling, running, etc.)

Exclusion Criteria:

* Intolerant to glucose (according to World Health Organization standards)
* Musculoskeletal injury or illness affecting exercise performance
* Failure to respect protocol guidelines (diet, exercise prior to experimentation, etc.)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive flexibility | Baseline (Before the exercise protocol), during the 3-minutes exercise bouts, and every 15 minutes during the 45 minutes following exercise.
  Measured with a computerized version of the 4th board of Stroop's Task.
Change in Mental Effort | Baseline (Before the exercise protocol), during the 3-minutes exercise bouts, and every 15 minutes during the 45 minutes following exercise.
  Measured with the DP-15 Scale, ranging from 1 to 15, 1 corresponds to "very, very easy" and 15 is "very, very hard"
Change in Perceived exertion | Baseline (Before the exercise protocol), during the 3-minutes exercise bouts, and every 15 minutes during the 45 minutes following exercise.
  Measured using a Category Ratio scale on 10 points (CR10), 0 signifies no exertion and 10 being maximal effort.
Change in Brain oxygenation | During Stroop's task (i.e.before the exercise protocol, during the 3-minutes exercise bouts, and every 15 minutes during the 45 minutes following exercise).
  Measured with near-infrared spectroscopy (NIRS).

SECONDARY OUTCOMES:
Change in Blood glucose concentration | Baseline (Before the exercise protocol), during the 3-minutes exercise bouts, and every 15 minutes during the 45 minutes following exercise.
  Measured by a puncture on the tip of the finger to collect a droplet of blood and process it with a commercial glucometer.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Tremblay, Principal Investigator — Associate Professor; Olivier Dupuy, Ph.D., Study Director — Professor
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada